CLINICAL TRIAL: NCT00345046
Title: A Comparison of Three Different Formulations of Topical Prednisolone Acetate 1% for Control of Post Glaucoma and/or Cataract Surgery Inflammation.
Brief Title: A Comparison of Three Different Formulations of Prednisolone Acetate 1%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0201-28
Record Dates: First submitted 2006-06-26; First posted 2006-06-27 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2014-03

CONDITIONS: Glaucoma; Cataract
Keywords: Glaucoma; Cataract
MeSH Terms: conditions — Glaucoma; Cataract | interventions — prednisolone acetate; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pred Forte 1% (Active Comparator): Pred Forte 1% dosed four times daily decreasing to once daily over four weeks.
  Interventions: Drug: Pred Forte
- EconoPred Plus 1% (Active Comparator): EconoPred Plus 1% dosed four times daily decreasing to once daily over four weeks.
  Interventions: Drug: EconoPred Plus
- Prednisolone Acetate 1% (Active Comparator): Prednisolone Acetate 1% dosed four times daily decreasing to once daily over four weeks.
  Interventions: Drug: Prednisolone Acetate

INTERVENTIONS:
Drug: Pred Forte — Four drops daily decreasing to once daily over four weeks.
  Other Names: Econopred Plus
  Arms: Pred Forte 1%
Drug: EconoPred Plus — Prednisolone Acetate four times daily decreasing to once daily over four weeks.
  Other Names: Pred Forte
  Arms: EconoPred Plus 1%
Drug: Prednisolone Acetate — Dosed four times daily decreasing to once daily over four weeks.
  Other Names: Pred Forte; EconoPred Plus
  Arms: Prednisolone Acetate 1%

SUMMARY:
Generic prednisolone acetate 1% is less effective than Pred Forte 1% or Econopred Plus 1%.

DETAILED DESCRIPTION:
Overall Study Design:

Structure:

This is a randomized, double-masked prospective study. The study medications will be masked and randomized by the outpatient pharmacy at Indiana University Hospital.

Duration:

Treatment duration: The duration of each subject's participation will be for up to 2 months after surgery. One hundred and two subjects will be enrolled over a twelve-month time span.

Controls:

Examiner, staff, and subjects are masked. Parallel group comparison.

Dosage/Dose Regimen/Instructions:

Subjects scheduled for glaucoma and/or cataract surgery will be recruited. Subjects may not be currently on any steroid or ophthalmic non-steroidal anti-inflammatory (NSAID) therapy for a minimum of 6 weeks prior to surgery. Subjects will be randomized to receive a dose of Pred Forte 1% (Allergan), Econopred Plus 1% (Alcon) or prednisolone acetate 1% (Falcon) four times a day starting immediately after finishing the surgery for two weeks, then twice a day for two more weeks. After 1 month of therapy subjects will stop or continue steroid treatment based on clinical findings. No other subconjunctival steroid or ointment will be used intra-operatively or post-operatively. The eye drop will be instilled per labeling instructions.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent.
* Be able and willing to follow instructions on the use of the study medication and likely to complete the entire course of the study.
* Be male or female of any race at least 18 years of age.
* Have visually significant cataract or medically uncontrolled glaucoma for which they have elected to undergo surgery.

Exclusion Criteria:

* Contraindication to use of corticosteroids.
* Ocular disease other than glaucoma or ocular hypertension that would interfere with study parameters (such as: uveitis, ocular infection, or severe dry eye). Subjects with mild chronic blepharitis, age-related macular degeneration and background diabetic retinopathy may be enrolled at the discretion of the investigator.
* Laser or any other intraocular surgery within the past three months.
* Require use of ocular NSAID or systemic steroids.
* Have known allergy or sensitivity to the study medications or their components
* Have corneal abnormalities that would interfere with the ability to obtain an adequate laser flare measurement.
* Be concurrently enrolled in an investigational drug or device study or participation within the last 30 days in any investigational drug or device study.
* Be pregnant, nursing, planning a pregnancy, or be of childbearing potential and not using a reliable form of contraception (a woman is considered of childbearing potential unless she is postmenopausal, has had a uterus and/or both ovaries removed, or has had a bilateral tubal ligation).
* Have a situation or condition that in the investigator's opinion may put the subject at significant risk, may confound the study results, or may interfere significantly with participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis B Cantor, MD, Principal Investigator — IUPUI/Clarian
Locations (1):
- IU Eye at Carmel, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Cantor LB. Ophthalmic generic drug approval process: implications for efficacy and safety. J Glaucoma. 1997 Oct;6(5):344-9. doi: 10.1097/00061198-199710000-00011. No abstract available. PMID 9327353
- [Background] Stoughton RB. Are generic formulations equivalent to trade name topical glucocorticoids? Arch Dermatol. 1987 Oct;123(10):1312-4. PMID 3662563
- [Background] Olsen EA. A double-blind controlled comparison of generic and trade-name topical steroids using the vasoconstriction assay. Arch Dermatol. 1991 Feb;127(2):197-201. PMID 1990984
- [Background] Casale TB, Azzam SM, Miller RE, Oren J. Demonstration of therapeutic equivalence of generic and innovator beclomethasone in seasonal allergic rhinitis. SAR Study Group. Ann Allergy Asthma Immunol. 1999 May;82(5):435-41. doi: 10.1016/s1081-1206(10)62717-2. PMID 10353573
- [Background] Nell H, Louw CM, Cyster H, Williams Z, Bardin PG, Joubert JR. Therapeutic equivalence study of two formulations (innovator v. generic) of beclomethasone dipropionate in adult asthmatic patients. S Afr Med J. 2001 Jan;91(1):51-6. PMID 11236299
- [Background] Apt L, Henrick A, Silverman LM. Patient compliance with use of topical ophthalmic corticosteroid suspensions. Am J Ophthalmol. 1979 Feb;87(2):210-4. doi: 10.1016/0002-9394(79)90145-4. No abstract available. PMID 434075
- [Background] Hille K, Hans J, Manderscheid T, Spang S, Ruprecht KW. [Laser flare in combined cataract and glaucoma surgery]. Ophthalmologe. 2001 Jan;98(1):47-53. doi: 10.1007/s003470170199. German. PMID 11220271
- [Background] Shah SM, Spalton DJ, Taylor JC. Correlations between laser flare measurements and anterior chamber protein concentrations. Invest Ophthalmol Vis Sci. 1992 Sep;33(10):2878-84. PMID 1526738
- [Background] Fiscella RG, Gutta R, Goldstein DB, Viana MAG. Comparison of PredForte Brand to generic Prednisolone acette and loteprednol etabonate (lotemax) in a Rabbit Model of Inflammation. American Academy of Ophthalmology 2001 Annual Meeting, Poster 73 Session 2001.
- See also: Electronic Orange Book — https://www.fda.gov/cder/ob/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period Feb 2005 - Jun 2008 Subjects were recruited from surgical schedule.
Pre-assignment Details: One subject was disqualified due to previous laser treatment. One subject did not receive study medication therefore was discontinued from study participation.
Groups:
- EconPred Plus 1%: EconoPred Plus 1% dosed four times daily decreasing to once daily over four weeks.
Period: Overall Study
Arm/Group | Pred Forte 1% | EconPred Plus 1% | Prednisolone Acetate 1%
Started | 18 | 22 | 16
Completed | 17 | 21 | 14
Not Completed | 1 | 1 | 2
Not completed — Protocol Violation | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Pred Forte: Pred Forte 1% dosed four times daily decreasing to once daily over four weeks.
  Pred Forte: Four drops daily decreasing to once daily over four weeks.
- EconoPred Plus: EconoPred Plus 1% dosed four times daily decreasing to once daily over four weeks.
  EconoPred Plus: Prednisolone Acetate four times daily decreasing to once daily over four weeks.
- Prednisolone Acetate: Prednisolone Acetate 1% dosed four times daily decreasing to once daily over four weeks.
  Prednisolone Acetate: Dosed four times daily decreasing to once daily over four weeks.
- Total: Total of all reporting groups
Arm/Group | Pred Forte | EconoPred Plus | Prednisolone Acetate | Total
Number analyzed (Participants) | 18 | 21 | 12 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (15.2) | 68.3 (13.0) | 65.7 (16.6) | 66.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 7 | 25
  Male | 8 | 13 | 5 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Flare at Resolution
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: Percent change in flare
Groups:
- Econo Pred Plus 1%: EconoPred Plus 1% dosed four times daily decreasing to once daily over four weeks.
  EconoPred Plus: Prednisolone Acetate four times daily decreasing to once daily over four weeks.
- Predisolone Acetate 1%: Prednisolone Acetate 1% dosed four times daily decreasing to once daily over four weeks.
  Prednisolone Acetate: Dosed four times daily decreasing to once daily over four weeks.
Arm/Group | Pred Forte 1% | Econo Pred Plus 1% | Predisolone Acetate 1%
Number analyzed (Participants) | 18 | 21 | 12
Percent change in flare | 64.8 (15.2) | 68.3 (13.0) | 65.7 (16.6)

ADVERSE EVENTS:
Arm/Group | Pred Forte 1% | EconoPred Plus 1% | Prednisolone Acetate 1%
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/21 | 0/12
Other Adverse Events (participants affected / at risk) | 0/18 | 0/21 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No